CLINICAL TRIAL: NCT02316470
Title: Dose Confirmation, Immunogenicity and Safety Study of the Clostridium Difficile Vaccine Candidate VLA84 in Healthy Adults Aged 50 Years and Older. Randomized, Controlled, Observer Blind Phase II Study
Brief Title: Dose-Confirmation, Immunogenicity and Safety Study of the Clostridium Difficile Vaccine Candidate VLA84 in Healthy Adults Aged 50 Years and Older. Phase II Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VLA84-201
Record Dates: First submitted 2014-12-09; First posted 2014-12-15 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-04

CONDITIONS: Clostridium Difficile
Keywords: Clostridium difficile; Valneva; Phase 2; Healthy adults

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- VLA84 75 mcg (microgram) w/o Alum (Active Comparator): VLA84 75 mcg w/o Alum consists of 0.75 mL (milliliters) VLA84 w/o Alum and 0.75 mL Placebo Vaccination Days: 0, 7 and 28 each with two injections
  Interventions: Biological: VLA84; Biological: Placebo
- VLA84 200 mcg w/o Alum (Active Comparator): VLA84 200 mcg w/o Alum consists of 2 injections each with 1.0 mL (milliliters) VLA84 w/o Alum Vaccination Days: 0, 7 and 28 each with two injections
  Interventions: Biological: VLA84
- VLA84 200 mcg with Alum (Active Comparator): VLA84 200 mcg with Alum consists of 2 injections each with 1.0 mL (milliliters) VLA84 with Alum Vaccination Days: 0, 7 and 28 each with two injections
  Interventions: Biological: VLA84
- Placebo (Placebo Comparator): Placebo consists of 2 injections each with 1.0 mL PBS (Phosphate Buffered Saline) Vaccination Days: 0, 7 and 28 each with two injections
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VLA84 — a recombinant fusion protein consisting of truncated Clostridium difficile (C. difficile) Toxin A and Toxin B
  Arms: VLA84 200 mcg w/o Alum; VLA84 200 mcg with Alum; VLA84 75 mcg (microgram) w/o Alum
Biological: Placebo — phosphate buffered saline (PBS) solution
  Arms: Placebo; VLA84 75 mcg (microgram) w/o Alum

SUMMARY:
Phase 2, randomized, observer-blind, placebo-controlled, multi-centric study including 4 parallel study groups.

500 Subjects (thereof, 250 aged 50 - 64 years and 250 aged 65 years and older) will be randomized in a (3:3:3:1) ratio to receive either VLA84 75 µg w/o (without) Alum, VLA84 200 µg w/o Alum, VLA84 200 µg w/ (with) Alum (150 subjects each), or placebo (50 subjects), as i.m. (intramuscular) vaccinations into alternating arms, on Days 0, 7 and 28

DETAILED DESCRIPTION:
This is a randomized, controlled, observer-blind Phase 2 study which aims to confirm the optimal dose and formulation of VLA84 in healthy adults aged ≥ 50 years of age. The study will be enrolled in two age strata, subjects aged 50 - 64 years and subjects aged 65 years and older, in a 1:1 ratio.

500 subjects (thereof, 250 aged 50 - 64 years and 250 aged 65 years and older) will be randomized in a 3:3:3:1 ratio to receive either VLA84 75 µg w/o Alum, VLA84 200 µg w/o Alum, VLA84 200 µg w/ Alum (150 subjects each), or placebo (50 subjects). Vaccinations consist of two i.m. injections administered in close proximity to each other in the deltoid region at Day 0, 7 and 28, starting with the non-dominant arm and alternating arms between the vaccination days.

The study will investigate the immunogenicity and safety of VLA84 up to six months after the last vaccination, i.e. 210 days per subject. The study includes eight outpatient visits on days 0, 7, 14, 28, 35, 56, 120 and 210. Serum will be collected to assess humoral immunity at days 0, 7, 14, 28, 35, 56, 120 and 210.

The study is OBSERVER blind. This means only pre-defined study staff will be unblinded, e.g., staff responsible for IMP accountability, preparation and administration, monitor responsible IMP accountability, or safety staff in case of safety reasons. All other persons involved in study conduct will remain blinded.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥50 years of good general health, including subjects with pharmacologically controlled conditions like hypercholesterolemia, hypertension, or type 2 diabetes mellitus.
* Informed consent form has been signed and dated

Exclusion Criteria:

* Subjects with any confirmed or suspected prior Clostridium difficile infection episode
* Previous vaccination against Clostridium difficile with any (investigational) vaccine or receipt of (investigational) monoclonal antibodies against Clostridium difficile toxins
* Use of any other investigational or non-registered medicinal product within 30 days prior to VLA84 vaccination at Visit 1 (Day 0) and throughout the entire study period.
* Active or passive vaccination four weeks before first vaccination at Visit 1 and during the entire study period, except for influenza (seasonal or pandemic) and pneumococcal vaccines which may be administered outside a 7-days interval before and after any trial vaccination
* Subject is pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year or surgically sterile)
* Known thrombocytopenia, bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion or until Visit 4 (Day28), contraindicating i.m. vaccination as judged by the investigator
* Clinically relevant renal, hepatic, cardiac, pulmonary or central nervous disorders, as judged by the investigator. Subjects with hypercholesterolemia, hypertension, or type 2 diabetes mellitus requiring medication are allowed if disease is adequately controlled
* Receipt of blood or blood-derived products in the past 3 months or anticipation of such products during the study period
* Known congenital, hereditary or acquired immunodeficiency, including known infection with human immunodeficiency virus (HIV), administration of chronic (defined as longer than 14 days) immunosuppressants or other immune-modifying drugs within 30 days prior to VLA84 vaccination at Visit 1 (Day 0) and during the study until Visit 5 (Day 35). For corticosteroids this means prednisone or equivalent ≥ 0.05 mg/kg/day; topical and inhaled steroids are allowed. Periodic steroid injections, e.g., intra-articular, are not allowed within 30 days prior to first VLA84 vaccination at Visit 1 (Day 0) and until Visit 5 (Day 35)
* History of autoimmune disease, including Type I Diabetes mellitus. Subjects with vitiligo or thyroid disease taking thyroid hormone replacement are not excluded
* Any malignancy in the past 5 years. If treatment for cancer was successfully completed more than 5 years ago and the malignancy is considered to be cured, the subject may be enrolled
* Known hypersensitivity or allergic reactions to one of the components of the vaccine
* Inability or unwillingness to provide informed consent
* Persons who are committed to an institution (by virtue of an order issued either by the judicial or the administrative authorities)
* Persons who are in a dependent relationship with the sponsor, an investigator or other study team members, or the study center. Dependent relationships include close relatives and household members (i.e., children, partner/spouse, siblings, parents) as well as employees of the investigator or study center personnel

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Dubischar, Study Director — Valneva Austria GmbH
Locations (10):
- United States (7):
  - Optimal Research LLC, Huntsville, Alabama
  - eStudy Site, Chula Vista, Chula Vista, California
  - eStudy Site, La Mesa, La Mesa, California
  - eStudy Site, Oceanside, Oceanside, California
  - Optimal Research LLC, Melbourne, Florida
  - Optimal Research LLC, Peoria, Illinois
  - Optimal Research LLC, Mishawaka, Indiana
- Germany (3):
  - Berliner Zentrum für Reise- und Tropenmedizin, Berlin
  - KFGN Klinische Forschung Hannover- Mitte GmbH, Hanover
  - Klinik und Poliklinik für Innere Medizin der Universität Rostock, Rostock

RESULTS

PARTICIPANT FLOW:
Groups:
- VLA84 75 mcg (Microgram) w/o Alum: VLA84 75 mcg w/o Alum consists of 1 injection of 0.75 mL (milliliters) VLA84 w/o Alum and 1 injection of 0.75 mL Placebo Vaccination Days: 0, 7 and 28
  VLA84: a recombinant fusion protein consisting of truncated Clostridium difficile (C. difficile) Toxin A and Toxin B
  Placebo: phosphate buffered saline (PBS) solution
- VLA84 200 mcg w/o Alum: VLA84 200 mcg w/o Alum consists of 2 injections each with 1.0 mL (milliliters) VLA84 w/o Alum Vaccination Days: 0, 7 and 28
  VLA84: a recombinant fusion protein consisting of truncated Clostridium difficile (C. difficile) Toxin A and Toxin B
- VLA84 200 mcg w/ Alum: VLA84 200 mcg w/ (with) Alum consists of 2 injections each with 1.0 mL (milliliters) VLA84 with Alum Vaccination Days: 0, 7 and 28
  VLA84: a recombinant fusion protein consisting of truncated Clostridium difficile (C. difficile) Toxin A and Toxin B
- Placebo: Placebo consists of 2 injections each with 1.0 mL PBS (Phosphate Buffered Saline) Vaccination Days: 0, 7 and 28
  Placebo: phosphate buffered saline (PBS) solution
Period: Overall Study
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg w/ Alum | Placebo
Started | 148 | 152 | 152 | 48
Completed | 143 | 146 | 147 | 46
Not Completed | 5 | 6 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo | Total
Number analyzed (Participants) | 148 | 152 | 152 | 48 | 500
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 72 | 77 | 77 | 24 | 250
  >=65 years | 76 | 75 | 75 | 24 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (8.86) | 64.1 (9.34) | 63.9 (9.15) | 63.7 (9.49) | 64.0 (9.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 82 | 87 | 24 | 268
  Male | 73 | 70 | 65 | 24 | 232
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 118 | 119 | 118 | 39 | 394
  Germany | 30 | 33 | 34 | 9 | 106

OUTCOME MEASURES:

1. Primary Outcome: Seroconversion Rate (SCR) on Day 56
Description: Seroconversion Rate (SCR), defined as percentage of subjects achieving a ≥4-fold increase in antibody titer from Day 0, for IgG against both Toxin A and Toxin B on Day 56;
Time Frame: Day 56
Population: per-protocol population,i.e., subjects who received at least one study vaccination without any major protocol deviation up to Day 210
Measure: Number (95% Confidence Interval); unit: percentage of study participants
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 137 | 135 | 141 | 46
percentage of study participants | 71.5 [63.5 to 78.4] | 83.0 [75.7 to 88.4] | 59.6 [51.3 to 67.3] | 0.0 [0.0 to 7.7]
Statistical Analysis 1: Comparison: VLA84 75 mcg (Microgram) w/o Alum vs VLA84 200 mcg w/o Alum vs VLA84 200 mcg With Alum vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: VLA84 75 mcg (Microgram) w/o Alum vs VLA84 200 mcg w/o Alum; Test type: Superiority or Other; p = 0.0261, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: VLA84 75 mcg (Microgram) w/o Alum vs VLA84 200 mcg With Alum; Test type: Superiority or Other; p = 0.0364, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: VLA84 75 mcg (Microgram) w/o Alum vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: VLA84 200 mcg w/o Alum vs VLA84 200 mcg With Alum; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: VLA84 200 mcg w/o Alum vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: VLA84 200 mcg With Alum vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

2. Secondary Outcome: SCR for IgG (Immunoglobulin G) Against Both Toxin A and Toxin B
Description: Seroconversion Rate (SCR), defined as percentage of subjects achieving a ≥4-fold increase in antibody titer from Day 0, for IgG against both Toxin A and Toxin B on Day 14, 28, 35, 120 and 210;
Time Frame: Days 14, 28, 35, 120 and 210
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 137 | 135 | 141 | 46
percentage of participants
  SCR at Day 14: number analyzed (Participants) | 137 | 134 | 141 | 46
  SCR at Day 14 | 31.4 [24.2 to 39.6] | 38.8 [31.0 to 47.3] | 27.7 [20.9 to 35.6] | 2.2 [0.4 to 11.3]
  SCR at Day 28 | 38.0 [30.3 to 46.3] | 49.6 [41.3 to 58.0] | 37.6 [30.0 to 45.8] | 2.2 [0.4 to 11.3]
  SCR at Day 35 | 56.9 [48.6 to 64.9] | 68.9 [60.6 to 76.1] | 50.4 [42.2 to 58.5] | 2.2 [0.4 to 11.3]
  SCR at Day 120: number analyzed (Participants) | 137 | 133 | 140 | 45
  SCR at Day 120 | 64.2 [55.9 to 71.8] | 77.4 [69.6 to 83.7] | 53.6 [45.3 to 61.1] | 0.0 [0.0 to 7.9]
  SCR at Day 210: number analyzed (Participants) | 134 | 132 | 137 | 45
  SCR at Day 210 | 54.5 [46.0 to 62.7] | 68.9 [60.6 to 76.2] | 44.5 [36.5 to 52.9] | 0.0 [0.0 to 7.9]
Statistical Analysis 1: Comparison: VLA84 75 mcg (Microgram) w/o Alum vs VLA84 200 mcg w/o Alum vs VLA84 200 mcg With Alum vs Placebo; statistical test was applied across all treatment groups at each of the listed time points; Test type: Superiority or Other; p < 0.0001, Fisher-Freeman-Halton Test — p-value was <0.0001 at each time point (Day 14, 28, 35, 120, 210)

3. Secondary Outcome: Seroconversion Rate (SCR) for IgG Against Toxin A
Description: Seroconversion Rate (SCR), defined as percentage of subjects achieving a ≥4-fold increase in antibody titer from Day 0, for IgG against Toxin A;
Time Frame: 14, 28, 35, 56, 120 and 210
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 137 | 135 | 141 | 46
percentage of participants
  SCR at Day 14: number analyzed (Participants) | 137 | 134 | 141 | 46
  SCR at Day 14 | 36.5 [28.9 to 44.8] | 46.3 [38.0 to 54.7] | 36.2 [28.7 to 44.4] | 4.3 [1.2 to 14.5]
  SCR at Day 28 | 51.8 [43.5 to 60.0] | 63.0 [54.6 to 70.6] | 69.5 [61.5 to 76.5] | 4.3 [1.2 to 14.5]
  SCR at Day 35 | 70.1 [61.9 to 77.1] | 80.0 [72.5 to 85.9] | 90.8 [84.9 to 94.5] | 4.3 [1.2 to 14.5]
  SCR at Day 56 | 92.0 [86.2 to 95.5] | 94.1 [88.7 to 97.0] | 96.5 [92.0 to 98.5] | 0.0 [0.0 to 7.7]
  SCR at Day 120: number analyzed (Participants) | 137 | 133 | 140 | 45
  SCR at Day 120 | 88.3 [81.9 to 92.7] | 91.7 [85.8 to 95.3] | 95.7 [91.0 to 98.0] | 0.0 [0.0 to 7.9]
  SCR at Day 210: number analyzed (Participants) | 134 | 132 | 137 | 45
  SCR at Day 210 | 85.1 [78.1 to 90.1] | 87.1 [80.3 to 91.8] | 93.4 [88.0 to 96.5] | 2.2 [0.4 to 11.6]
Statistical Analysis 1: Comparison: VLA84 75 mcg (Microgram) w/o Alum vs VLA84 200 mcg w/o Alum vs VLA84 200 mcg With Alum vs Placebo; statistical test was applied across all treatment groups at each of the listed time points; Test type: Superiority or Other; p < 0.0001, Fisher-Freeman-Halton Test — p-value was <0.0001 at each time point (Day 14, 28, 35, 56, 120, 210)

4. Secondary Outcome: Seroconversion Rate (SCR) for IgG Against Toxin B
Description: Seroconversion Rate (SCR), defined as percentage of subjects achieving a ≥4-fold increase in antibody titer from Day 0, for IgG against Toxin B;
Time Frame: Days 14, 28, 35, 56, 120 and 210
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 137 | 135 | 141 | 46
percentage of participants
  SCR at Day 14: number analyzed (Participants) | 137 | 134 | 141 | 46
  SCR at Day 14 | 35.0 [27.6 to 43.3] | 44.0 [35.9 to 52.5] | 35.5 [28.0 to 43.6] | 2.2 [0.4 to 11.3]
  SCR at Day 28 | 41.6 [33.7 to 50.5] | 53.3 [44.9 to 61.5] | 41.1 [33.4 to 49.4] | 2.2 [0.4 to 11.3]
  SCR at Day 35 | 56.9 [48.6 to 64.9] | 70.4 [62.2 to 77.4] | 50.4 [42.2 to 58.5] | 4.3 [1.2 to 14.5]
  SCR at Day 56 | 71.5 [63.5 to 78.4] | 83.7 [76.6 to 89.0] | 59.6 [51.3 to 67.3] | 2.2 [0.4 to 11.3]
  SCR at Day 120: number analyzed (Participants) | 137 | 133 | 140 | 45
  SCR at Day 120 | 64.2 [55.9 to 71.8] | 78.2 [70.4 to 84.4] | 54.3 [46.0 to 62.3] | 0.0 [0.0 to 7.9]
  SCR at Day 210: number analyzed (Participants) | 134 | 132 | 137 | 45
  SCR at Day 210 | 55.2 [46.8 to 63.4] | 70.5 [62.2 to 77.6] | 45.3 [37.2 to 53.6] | 0.0 [0.0 to 7.9]
Statistical Analysis 1: Comparison: VLA84 75 mcg (Microgram) w/o Alum vs VLA84 200 mcg w/o Alum vs VLA84 200 mcg With Alum vs Placebo; statistical test was applied across all treatment groups at each of the listed time points; Test type: Superiority or Other; p < 0.0001, Fisher-Freeman-Halton Test — the p-value was <0.0001 at each time point (Day 14, 28, 35, 56, 120, 210)

5. Secondary Outcome: Geometric Mean Titer (GMT) for IgG Against Toxin A
Description: Geometric Mean Titer (GMT) for IgG against Toxin A as determined by ELISA on Days 0, 14, 28, 35, 56 (primary endpoint time point), 120 and 210;
Time Frame: Days 0, 14, 28, 35, 56, 120 and 210
Population: PP210 = per protocol population defined as subjects without major protocol deviation up to Day 210
Measure: Geometric Mean (95% Confidence Interval); unit: EU/ml
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 137 | 135 | 141 | 46
EU/ml
  GMT at Day 0 | 40.5 [35.7 to 45.9] | 37.4 [33.4 to 41.8] | 44.9 [39.2 to 51.4] | 37.6 [30.0 to 47.2]
  GMT at Day 14: number analyzed (Participants) | 137 | 134 | 141 | 46
  GMT at Day 14 | 227.2 [144.4 to 357.6] | 350.9 [216.6 to 568.4] | 226.1 [144.9 to 352.6] | 38.1 [29.4 to 49.3]
  GMT at Day 28 | 412.3 [266.4 to 638.1] | 623.2 [398.2 to 975.3] | 717.7 [495.7 to 1039.1] | 36.3 [28.4 to 46.6]
  GMT at Day 35 | 1056.6 [680.4 to 1640.9] | 2083.7 [1370.8 to 3167.3] | 3545.6 [2577.4 to 4877.6] | 34.9 [28.1 to 43.3]
  GMT at Day 56 | 2868.9 [2068.9 to 3978.1] | 4328.5 [3160.5 to 5928.3] | 4687.6 [3650.6 to 6019.3] | 33.9 [28.4 to 40.3]
  GMT at Day 120: number analyzed (Participants) | 137 | 133 | 140 | 45
  GMT at Day 120 | 1563.5 [1157.2 to 2112.6] | 2533.8 [1867.4 to 3438.0] | 2416.7 [1926.7 to 3031.3] | 31.4 [27.1 to 36.4]
  GMT at Day 210: number analyzed (Participants) | 134 | 132 | 137 | 45
  GMT at Day 210 | 866.0 [650.1 to 1153.6] | 1395.3 [1044.1 to 1864.7] | 1288.8 [1037.9 to 1600.5] | 34.3 [27.7 to 42.5]

6. Secondary Outcome: Geometric Mean Titer (GMT) for IgG Against Toxin B
Description: Geometric Mean Titer (GMT) for IgG against Toxin B as determined by ELISA on Days 0, 14, 28, 35, 56 (primary endpoint time point), 120 and 210;
Time Frame: Days 0, 14, 28, 35, 56, 120 and 210
Population: PP210 = per protocol population defined as subjects without major protocol deviation up to Day 210
Measure: Geometric Mean (95% Confidence Interval); unit: EU/ml
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 137 | 135 | 141 | 46
EU/ml
  GMT at Day 0 | 150.1 [126.2 to 178.5] | 107.4 [90.3 to 127.8] | 131.9 [109.0 to 159.6] | 104.3 [73.6 to 147.7]
  GMT at Day 14: number analyzed (Participants) | 137 | 134 | 141 | 46
  GMT at Day 14 | 778.4 [478.7 to 1265.8] | 951.8 [561.1 to 1614.6] | 585.0 [359.7 to 951.6] | 98.8 [69.4 to 140.7]
  GMT at Day 28 | 949.2 [602.3 to 1495.9] | 1026.5 [636.2 to 1656.2] | 754.5 [476.3 to 1195.2] | 107.6 [76.8 to 150.7]
  GMT at Day 35 | 1651.4 [1070.3 to 2547.9] | 2377.1 [1558.6 to 3625.4] | 1165.9 [763.4 to 1780.9] | 107.0 [75.3 to 151.9]
  GMT at Day 56 | 2370.5 [1641.2 to 3423.8] | 3336.5 [2398.9 to 4640.7] | 1449.4 [1001.8 to 2097.2] | 107.8 [77.0 to 151.0]
  GMT at Day 120: number analyzed (Participants) | 137 | 133 | 140 | 45
  GMT at Day 120 | 1304.5 [942.0 to 1806.5] | 1699.9 [1250.0 to 2311.6] | 881.3 [632.1 to 1228.8] | 92.1 [66.1 to 128.2]
  GMT at Day 210: number analyzed (Participants) | 134 | 132 | 137 | 45
  GMT at Day 210 | 863.3 [639.8 to 1165.0] | 1023.0 [770.8 to 1357.7] | 595.4 [431.7 to 821.1] | 96.1 [69.1 to 133.5]

7. Secondary Outcome: GMT for Toxin A Neutralizing Antibodies
Description: GMT for Toxin A neutralizing antibodies (TNA) as determined by Toxin Neutralization Assay on Days 0, 35, 56, 120* and 210
  * TNA in sera from Day 120 were to be measured only if meaningful in view of the Day 56 and Day 210 results; in fact Day 120 TNA was not measured.
Time Frame: Days 0, 35, 56, 120 and 210
Population: PP210 = per protocol population defined as subjects without major protocol deviation up to Day 210
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 137 | 135 | 141 | 46
Titer
  GMT at Day 0 | 11.0 [10.2 to 11.8] | 10.3 [9.9 to 10.8] | 10.8 [10.1 to 11.5] | 10.0 [10.0 to 10.0]
  GMT at Day 35 | 93.5 [63.3 to 138.1] | 155.2 [104.9 to 229.7] | 148.7 [104.3 to 211.9] | 10.3 [9.7 to 10.9]
  GMT at Day 56 | 143.1 [102.4 to 200.0] | 200.9 [144.1 to 280.0] | 153.3 [112.5 to 209.0] | 10.3 [9.9 to 10.9]
  GMT at Day 210: number analyzed (Participants) | 134 | 132 | 137 | 45
  GMT at Day 210 | 95.1 [69.2 to 130.7] | 168.7 [122.6 to 232.3] | 189.4 [148.1 to 242.3] | 10.2 [9.8 to 10.6]

8. Secondary Outcome: GMT for Toxin B Neutralizing Antibodies
Description: GMT for Toxin B neutralizing antibodies (TNA) as determined by Toxin Neutralization Assay on Days 0, 35, 56, 120* and 210
  * TNA in sera from Day 120 were to be measured only if meaningful in view of the Day 56 and Day 210 results; in fact Day 120 TNA was not measured.
Time Frame: Days 0, 35, 56, 120 and 210
Population: PP210 = per protocol population defined as subjects without major protocol deviation up to Day 210
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 137 | 135 | 141 | 46
Titer
  GMT at Day 0 | 17.4 [14.4 to 20.9] | 15.9 [13.5 to 18.8] | 19.1 [15.5 to 23.6] | 18.3 [13.0 to 25.7]
  GMT at Day 35 | 72.9 [51.0 to 104.3] | 99.6 [71.0 to 139.9] | 61.6 [44.0 to 86.4] | 18.6 [13.3 to 26.1]
  GMT at Day 56 | 69.8 [50.8 to 95.9] | 74.3 [55.4 to 99.6] | 52.3 [38.4 to 71.1] | 19.1 [13.9 to 26.2]
  GMT at Day 210: number analyzed (Participants) | 134 | 132 | 137 | 45
  GMT at Day 210 | 51.0 [37.9 to 68.8] | 61.0 [46.3 to 80.4] | 43.0 [31.7 to 58.3] | 17.2 [12.5 to 23.7]

9. Secondary Outcome: SCR for IgG Against Toxin A, Against Toxin B and Against Both Toxin A and Toxin B Stratified by Age Group
Description: Seroconversion Rate (SCR) for IgG against Toxin A, against Toxin B and against both Toxin A and Toxin B on Days 14, 28, 35, 56, 120 and 210, stratified by age group (subjects 50 - < 65 years and 65 years and older)
Time Frame: Days 14, 28, 35, 56, 120 and 210
Population: PP210 = per protocol population defined as subjects without major protocol deviation up to Day 210
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 137 | 135 | 141 | 46
percentage of participants
  SCR against Toxin A and B at Day 14; 50 to < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  SCR against Toxin A and B at Day 14; 50 to < 65 | 31.3 [21.5 to 43.2] | 42.6 [31.6 to 54.5] | 27.1 [18.1 to 38.5] | 4.5 [0.8 to 21.8]
  SCR against Toxin A and B at Day 28; 50 to < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  SCR against Toxin A and B at Day 28; 50 to < 65 | 32.8 [22.8 to 44.7] | 54.4 [42.7 to 65.7] | 34.3 [24.2 to 46.0] | 4.5 [0.8 to 21.8]
  SCR against Toxin A and B at Day 35; 50 to < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  SCR against Toxin A and B at Day 35; 50 to < 65 | 55.2 [43.4 to 66.5] | 72.1 [60.4 to 81.3] | 50.0 [38.6 to 61.4] | 4.5 [0.8 to 21.8]
  SCR against Toxin A and B at Day 56; 50 to < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  SCR against Toxin A and B at Day 56; 50 to < 65 | 70.1 [58.3 to 79.8] | 86.8 [76.7 to 92.9] | 60.0 [48.3 to 70.7] | 0.0 [0.0 to 14.9]
  SCR against Toxin A and B at Day 120; 50 to < 65: number analyzed (Participants) | 67 | 67 | 70 | 22
  SCR against Toxin A and B at Day 120; 50 to < 65 | 58.2 [46.3 to 69.3] | 80.6 [69.6 to 88.3] | 50.0 [38.6 to 61.4] | 0.0 [0.0 to 14.9]
  SCR against Toxin A and B at Day 210; 50 to < 65: number analyzed (Participants) | 65 | 66 | 68 | 22
  SCR against Toxin A and B at Day 210; 50 to < 65 | 47.7 [36.0 to 59.6] | 72.7 [61.0 to 82.0] | 41.2 [30.3 to 53.0] | 0.0 [0.0 to 14.9]
  SCR against Toxin A and B at Day 14; 65 and older: number analyzed (Participants) | 70 | 66 | 71 | 24
  SCR against Toxin A and B at Day 14; 65 and older | 31.4 [21.8 to 43.0] | 34.8 [24.5 to 46.9] | 28.2 [19.0 to 39.5] | 0.0 [0.0 to 13.8]
  SCR against Toxin A and B at Day 28; 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  SCR against Toxin A and B at Day 28; 65 and older | 42.9 [31.9 to 54.5] | 44.8 [33.5 to 56.6] | 40.8 [30.2 to 52.5] | 0.0 [0.0 to 13.8]
  SCR against Toxin A and B at Day 35; 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  SCR against Toxin A and B at Day 35; 65 and older | 58.6 [46.9 to 69.4] | 65.7 [53.7 to 75.9] | 50.7 [39.3 to 62.0] | 0.0 [0.0 to 13.8]
  SCR against Toxin A and B at Day 56; 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  SCR against Toxin A and B at Day 56; 65 and older | 72.9 [61.5 to 81.9] | 79.1 [67.9 to 87.1] | 59.2 [47.5 to 69.8] | 0.0 [0.0 to 13.8]
  SCR against Toxin A and B at Day 120; 65 and older: number analyzed (Participants) | 70 | 66 | 70 | 23
  SCR against Toxin A and B at Day 120; 65 and older | 70.0 [58.5 to 79.5] | 74.2 [62.6 to 83.3] | 57.1 [45.5 to 68.1] | 0.0 [0.0 to 14.3]
  SCR against Toxin A and B at Day 210; 65 and older: number analyzed (Participants) | 69 | 66 | 69 | 23
  SCR against Toxin A and B at Day 210; 65 and older | 60.9 [49.1 to 71.5] | 65.2 [53.1 to 75.5] | 47.8 [36.5 to 59.4] | 0.0 [0.0 to 14.3]
  SCR against Toxin A at Day 14; 50 to < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  SCR against Toxin A at Day 14; 50 to < 65 | 34.3 [24.1 to 46.3] | 52.9 [41.2 to 64.3] | 38.6 [28.0 to 50.3] | 9.1 [2.5 to 27.8]
  SCR against Toxin A at Day 28; 50 to < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  SCR against Toxin A at Day 28; 50 to < 65 | 49.3 [37.7 to 60.9] | 67.6 [55.8 to 77.6] | 74.3 [63.0 to 83.1] | 9.1 [2.5 to 27.8]
  SCR against Toxin A at Day 35; 50 to < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  SCR against Toxin A at Day 35; 50 to < 65 | 74.6 [63.1 to 83.5] | 85.3 [75.0 to 91.8] | 94.3 [86.2 to 97.8] | 9.1 [2.5 to 27.8]
  SCR against Toxin A at Day 56; 50 to < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  SCR against Toxin A at Day 56; 50 to < 65 | 89.6 [80.0 to 94.8] | 97.1 [89.9 to 99.2] | 95.7 [88.1 to 98.5] | 0.0 [0.0 to 14.9]
  SCR against Toxin A at Day 120; 50 to < 65: number analyzed (Participants) | 67 | 67 | 70 | 22
  SCR against Toxin A at Day 120; 50 to < 65 | 86.6 [76.4 to 92.8] | 94.0 [85.6 to 97.7] | 95.7 [88.1 to 98.5] | 0.0 [0.0 to 14.9]
  SCR against Toxin A at Day 210; 50 to < 65: number analyzed (Participants) | 65 | 66 | 68 | 22
  SCR against Toxin A at Day 210; 50 to < 65 | 81.5 [70.4 to 89.1] | 92.4 [83.5 to 96.7] | 95.6 [87.8 to 98.5] | 4.5 [0.8 to 21.8]
  SCR against Toxin A at Day 14; 65 and older: number analyzed (Participants) | 70 | 66 | 71 | 24
  SCR against Toxin A at Day 14; 65 and older | 38.6 [28.0 to 50.3] | 39.4 [28.5 to 51.5] | 33.8 [23.9 to 45.4] | 0.0 [0.0 to 13.8]
  SCR against Toxin A at Day 28; 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  SCR against Toxin A at Day 28; 65 and older | 54.3 [42.7 to 65.4] | 58.2 [46.3 to 69.3] | 64.8 [53.2 to 74.9] | 0.0 [0.0 to 13.8]
  SCR against Toxin A at Day 35; 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  SCR against Toxin A at Day 35; 65 and older | 65.7 [54.0 to 75.8] | 74.6 [63.1 to 83.5] | 87.3 [77.6 to 93.2] | 0.0 [0.0 to 13.8]
  SCR against Toxin A at Day 56; 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  SCR against Toxin A at Day 56; 65 and older | 94.3 [86.2 to 97.8] | 91.0 [81.8 to 95.8] | 97.2 [90.3 to 99.2] | 0.0 [0.0 to 13.8]
  SCR against Toxin A at Day 120; 65 and older: number analyzed (Participants) | 70 | 66 | 70 | 23
  SCR against Toxin A at Day 120; 65 and older | 90.0 [80.8 to 95.1] | 89.4 [79.7 to 94.8] | 95.7 [88.1 to 98.5] | 0.0 [0.0 to 14.3]
  SCR against Toxin A at Day 210; 65 and older: number analyzed (Participants) | 69 | 66 | 69 | 23
  SCR against Toxin A at Day 210; 65 and older | 88.4 [78.8 to 94.0] | 81.8 [70.9 to 89.3] | 91.3 [82.3 to 96.0] | 0.0 [0.0 to 14.3]
  SCR against Toxin B at Day 14; 50 to < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  SCR against Toxin B at Day 14; 50 to < 65 | 32.8 [22.8 to 44.7] | 45.6 [34.3 to 57.3] | 30.0 [20.5 to 41.5] | 4.5 [0.8 to 21.8]
  SCR against Toxin B at Day 28; 50 to < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  SCR against Toxin B at Day 28; 50 to < 65 | 37.3 [26.7 to 49.3] | 55.9 [44.1 to 67.1] | 35.7 [25.5 to 47.4] | 4.5 [0.8 to 21.8]
  SCR against Toxin B at Day 35; 50 to < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  SCR against Toxin B at Day 35; 50 to < 65 | 55.2 [43.4 to 66.5] | 72.1 [60.4 to 81.3] | 50.0 [38.6 to 61.4] | 9.1 [2.5 to 27.8]
  SCR against Toxin B at Day 56; 50 to < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  SCR against Toxin B at Day 56; 50 to < 65 | 70.1 [58.3 to 79.8] | 86.8 [76.7 to 92.9] | 60.0 [48.3 to 70.7] | 0.0 [0.0 to 14.9]
  SCR against Toxin B at Day 120; 50 to < 65: number analyzed (Participants) | 67 | 67 | 70 | 22
  SCR against Toxin B at Day 120; 50 to < 65 | 58.2 [46.3 to 69.3] | 80.6 [69.6 to 88.3] | 50.0 [38.6 to 61.4] | 0.0 [0.0 to 14.9]
  SCR against Toxin B at Day 210; 50 to < 65: number analyzed (Participants) | 65 | 66 | 68 | 22
  SCR against Toxin B at Day 210; 50 to < 65 | 49.2 [37.5 to 61.1] | 74.2 [62.6 to 83.3] | 41.2 [30.3 to 53.0] | 0.0 [0.0 to 14.9]
  SCR against Toxin B at Day 14; 65 and older: number analyzed (Participants) | 70 | 66 | 71 | 24
  SCR against Toxin B at Day 14; 65 and older | 37.1 [26.8 to 48.9] | 42.4 [31.2 to 54.4] | 40.8 [30.2 to 52.5] | 0.0 [0.0 to 13.8]
  SCR against Toxin B at Day 28; 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  SCR against Toxin B at Day 28; 65 and older | 45.7 [34.6 to 57.3] | 50.7 [39.1 to 62.3] | 46.5 [35.4 to 58.0] | 0.0 [0.0 to 13.8]
  SCR against Toxin B at Day 35; 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  SCR against Toxin B at Day 35; 65 and older | 58.6 [46.9 to 69.4] | 68.7 [56.8 to 78.5] | 50.7 [39.3 to 62.0] | 0.0 [0.0 to 13.8]
  SCR against Toxin B at Day 56; 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  SCR against Toxin B at Day 56; 65 and older | 72.9 [61.5 to 81.9] | 80.6 [69.6 to 88.3] | 59.2 [47.5 to 69.8] | 4.2 [0.7 to 20.2]
  SCR against Toxin B at Day 120; 65 and older: number analyzed (Participants) | 70 | 66 | 70 | 23
  SCR against Toxin B at Day 120; 65 and older | 70.0 [58.5 to 79.5] | 75.8 [64.2 to 84.5] | 58.6 [46.9 to 69.4] | 0.0 [0.0 to 14.3]
  SCR against Toxin B at Day 210; 65 and older: number analyzed (Participants) | 69 | 66 | 69 | 23
  SCR against Toxin B at Day 210; 65 and older | 60.9 [49.1 to 71.5] | 66.7 [54.7 to 76.8] | 49.3 [37.8 to 60.8] | 0.0 [0.0 to 14.3]

10. Secondary Outcome: GMT for IgG Against Toxin A and Against Toxin B Stratified by Age Group
Description: GMT for IgG against Toxin A and against Toxin B on Days 0, 14, 28, 35, 56, 120 and 210, stratified by age group (subjects 50 - < 65 years and 65 years and older)
Time Frame: Days 0, 14, 28, 35, 56, 120, 210
Population: PP210 = per protocol population defined as subjects without major protocol deviation up to Day 210
Measure: Geometric Mean (95% Confidence Interval); unit: EU/ml
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 137 | 135 | 141 | 46
EU/ml
  Toxin A: GMT at Day 0, 50 - < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  Toxin A: GMT at Day 0, 50 - < 65 | 42.6 [35.6 to 51.0] | 37.7 [32.4 to 43.9] | 41.2 [34.5 to 49.3] | 31.4 [2.45 to 40.3]
  Toxin A: GMT at Day 14, 50 - < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  Toxin A: GMT at Day 14, 50 - < 65 | 248.0 [126.1 to 487.7] | 531.3 [252.6 to 1117.5] | 216.4 [117.8 to 397.6] | 37.7 [25.6 to 55.7]
  Toxin A: GMT at Day 28, 50 - < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  Toxin A: GMT at Day 28, 50 - < 65 | 400.1 [213.3 to 750.3] | 851.8 [436.4 to 1662.5] | 704.2 [429.0 to 1155.7] | 37.1 [25.6 to 53.7]
  Toxin A: GMT at Day 35, 50 - < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  Toxin A: GMT at Day 35, 50 - < 65 | 1053.1 [562.9 to 1970.1] | 2579.7 [1444.9 to 4605.9] | 3502.1 [2274.0 to 5393.3] | 38.1 [25.4 to 57.1]
  Toxin A: GMT at Day 56, 50 - < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  Toxin A: GMT at Day 56, 50 - < 65 | 2581.7 [1642.1 to 4058.7] | 4566.4 [3027.4 to 6887.7] | 4344.8 [3077.1 to 6134.8] | 30.5 [23.6 to 39.5]
  Toxin A: GMT at Day 120, 50 - < 65: number analyzed (Participants) | 67 | 67 | 70 | 22
  Toxin A: GMT at Day 120, 50 - < 65 | 1391.8 [910.6 to 2127.3] | 2589.3 [1720.9 to 3896.0] | 2221.4 [1620.5 to 3045.0] | 29.9 [24.0 to 37.3]
  Toxin A: GMT at Day 210, 50 - < 65: number analyzed (Participants) | 65 | 66 | 68 | 22
  Toxin A: GMT at Day 210, 50 - < 65 | 792.9 [526.2 to 1194.8] | 1510.9 [1042.1 to 2190.7] | 1269.8 [921.6 to 1749.7] | 33.0 [24.7 to 44.2]
  Toxin A: GMT at Day 0, 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  Toxin A: GMT at Day 0, 65 and older | 38.5 [32.3 to 46.0] | 37.0 [31.3 to 43.8] | 48.8 [39.7 to 59.9] | 44.3 [30.4 to 64.6]
  Toxin A: GMT at Day 14, 65 and older: number analyzed (Participants) | 70 | 66 | 71 | 24
  Toxin A: GMT at Day 14, 65 and older | 209.0 [112.1 to 389.7] | 228.8 [124.0 to 422.3] | 236.0 [121.7 to 457.9] | 38.5 [26.5 to 55.8]
  Toxin A: GMT at Day 28, 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  Toxin A: GMT at Day 28, 65 and older | 424.4 [227.8 to 790.7] | 453.8 [248.4 to 829.1] | 731.4 [417.2 to 1282.0] | 35.6 [24.8 to 51.1]
  Toxin A: GMT at Day 35, 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  Toxin A: GMT at Day 35, 65 and older | 1060.0 [562.3 to 1998.3] | 1677.7 [906.5 to 3104.9] | 3589.1 [2221.7 to 5798.0] | 32.1 [25.8 to 40.1]
  Toxin A: GMT at Day 56, 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  Toxin A: GMT at Day 56, 65 and older | 3173.6 [1962.2 to 5133.0] | 4099.8 [2517.4 to 6676.7] | 5052.1 [3491.8 to 7309.7] | 37.3 [29.0 to 47.9]
  Toxin A: GMT at Day 120, 65 and older: number analyzed (Participants) | 70 | 66 | 70 | 23
  Toxin A: GMT at Day 120, 65 and older | 1747.7 [1130.8 to 2701.3] | 2478.7 [1556.9 to 3946.1] | 2629.1 [1886.1 to 3664.9] | 32.9 [26.6 to 40.7]
  Toxin A: GMT at Day 210, 65 and older: number analyzed (Participants) | 69 | 66 | 69 | 23
  Toxin A: GMT at Day 210, 65 and older | 941.1 [624.4 to 1418.4] | 1288.6 [817.9 to 2030.1] | 1307.8 [969.1 to 1765.0] | 35.6 [25.5 to 49.8]
  Toxin B: GMT at Day 0, 50 - < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  Toxin B: GMT at Day 0, 50 - < 65 | 142.6 [113.2 to 179.7] | 114.6 [91.8 to 142.9] | 131.7 [100.5 to 172.7] | 87.8 [57.4 to 134.4]
  Toxin B: GMT at Day 14, 50 - < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  Toxin B: GMT at Day 14, 50 - < 65 | 630.3 [323.6 to 1227.8] | 1101.1 [523.3 to 2316.7] | 476.7 [233.6 to 973.0] | 83.9 [54.6 to 128.7]
  Toxin B: GMT at Day 28, 50 - < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  Toxin B: GMT at Day 28, 50 - < 65 | 729.3 [391.8 to 1357.8] | 1292.3 [672.1 to 2484.8] | 569.8 [299.4 to 1084.6] | 94.8 [62.0 to 145.2]
  Toxin B: GMT at Day 35, 50 - < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  Toxin B: GMT at Day 35, 50 - < 65 | 1392.2 [759.2 to 2553.0] | 2962.2 [1677.0 to 5232.3] | 1039.7 [578.9 to 1867.3] | 103.3 [65.4 to 163.1]
  Toxin B: GMT at Day 56, 50 - < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  Toxin B: GMT at Day 56, 50 - < 65 | 1832.7 [1111.0 to 3023.2] | 3960.3 [2546.8 to 6158.5] | 1316.9 [777.9 to 2229.3] | 83.7 [53.9 to 130.1]
  Toxin B: GMT at Day 120, 50 - < 65: number analyzed (Participants) | 67 | 67 | 70 | 22
  Toxin B: GMT at Day 120, 50 - < 65 | 1034.5 [659.6 to 1622.4] | 2135.4 [1408.7 to 3237.0] | 745.6 [465.6 to 1193.8] | 79.7 [53.0 to 119.9]
  Toxin B: GMT at Day 210, 50 - < 65: number analyzed (Participants) | 65 | 66 | 68 | 22
  Toxin B: GMT at Day 210, 50 - < 65 | 714.1 [467.8 to 1090.1] | 1317.8 [894.2 to 1942.2] | 501.1 [314.3 to 799.0] | 79.2 [52.6 to 119.3]
  Toxin B: GMT at Day 0, 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  Toxin B: GMT at Day 0, 65 and older | 157.6 [121.3 to 204.8] | 100.6 [76.6 to 132.2] | 132.1 [100.3 to 174.0] | 122.1 [69.3 to 215.0]
  Toxin B: GMT at Day 14, 65 and older: number analyzed (Participants) | 70 | 66 | 71 | 24
  Toxin B: GMT at Day 14, 65 and older | 952.7 [464.3 to 1955.0] | 819.1 [379.5 to 1768.1] | 715.9 [364.0 to 1408.0] | 114.8 [64.5 to 204.5]
  Toxin B: GMT at Day 28, 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  Toxin B: GMT at Day 28, 65 and older | 1221.5 [623.7 to 2392.2] | 812.5 [398.7 to 1656.0] | 995.1 [511.1 to 1937.6] | 120.7 [70.2 to 207.6]
  Toxin B: GMT at Day 35, 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  Toxin B: GMT at Day 35, 65 and older | 1944.5 [1033.9 to 3657.3] | 1901.3 [1007.7 to 3587.3] | 1305.4 [698.7 to 2439.0] | 110.4 [63.1 to 193.1]
  Toxin B: GMT at Day 56, 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  Toxin B: GMT at Day 56, 65 and older | 3032.4 [1762.3 to 5217.7] | 2803.8 [1701.9 to 4619.1] | 1593.2 [937.3 to 2707.9] | 136.0 [81.1 to 227.9]
  Toxin B: GMT at Day 120, 65 and older: number analyzed (Participants) | 70 | 66 | 70 | 23
  Toxin B: GMT at Day 120, 65 and older | 1628.7 [1013.3 to 2617.7] | 1348.5 [853.6 to 2130.3] | 1041.9 [646.2 to 1679.8] | 105.7 [61.4 to 181.9]
  Toxin B: GMT at Day 210, 65 and older: number analyzed (Participants) | 69 | 66 | 69 | 23
  Toxin B: GMT at Day 210, 65 and older | 1032.3 [671.4 to 1587.3] | 794.1 [525.2 to 1200.7] | 705.6 [449.6 to 1107.4] | 115.5 [67.9 to 196.6]

11. Secondary Outcome: GMTs for Toxin A Neutralizing Antibodies and for Toxin B Neutralizing Antibodies Stratified by Age Group
Description: GMTs for Toxin A neutralizing antibodies and for Toxin B neutralizing antibodies as determined by Toxin Neutralization Assay on Days 0, 35, 56, 120* and 210, stratified by age group (subjects 50 - < 65 years and 65 years and older)
  * TNA in sera from Day 120 were to be measured only if meaningful in view of the Day 56 and Day 210 results; in fact Day 120 TNA was not measured.
Time Frame: Days 0, 35, 56, 120 and 210
Population: PP210 = per protocol population defined as subjects without major protocol deviation up to Day 210
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 137 | 135 | 141 | 46
Titer
  Toxin A: GMT at Day 0, 50 - < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  Toxin A: GMT at Day 0, 50 - < 65 | 10.8 [10.0 to 11.6] | 10.6 [9.7 to 11.6] | 10.9 [10.0 to 12.0] | 10.0 [10.0 to 10.0]
  Toxin A: GMT at Day 35, 50 - < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  Toxin A: GMT at Day 35, 50 - < 65 | 101.7 [56.0 to 184.5] | 199.4 [112.5 to 353.4] | 130.3 [82.4 to 206.1] | 10.6 [9.4 to 12.0]
  Toxin A: GMT at Day 56, 50 - < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  Toxin A: GMT at Day 56, 50 - < 65 | 138.2 [82.9 to 230.4] | 215.3 [130.5 to 355.1] | 124.3 [81.6 to 189.3] | 10.0 [10.0 to 10.0]
  Toxin A: GMT at Day 210, 50 - < 65: number analyzed (Participants) | 65 | 66 | 68 | 22
  Toxin A: GMT at Day 210, 50 - < 65 | 81.3 [49.9 to 132.4] | 187.5 [118.1 to 297.7] | 188.4 [135.1 to 262.6] | 10.0 [10.0 to 10.0]
  Toxin A: GMT at Day 0, 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  Toxin A: GMT at Day 0, 65 and older | 11.2 [9.8 to 12.7] | 10.0 [10.0 to 10.0] | 10.6 [9.6 to 11.6] | 10.0 [10.0 to 10.0]
  Toxin A: GMT at Day 35, 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  Toxin A: GMT at Day 35, 65 and older | 86.2 [51.2 to 145.3] | 120.4 [70.0 to 207.1] | 169.3 [97.8 to 293.1] | 10.0 [10.0 to 10.0]
  Toxin A: GMT at Day 56, 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  Toxin A: GMT at Day 56, 65 and older | 148.0 [94.5 to 231.6] | 187.3 [119.6 to 293.2] | 188.5 [119.0 to 298.6] | 10.7 [9.7 to 11.7]
  Toxin A: GMT at Day 210, 65 and older: number analyzed (Participants) | 69 | 66 | 69 | 23
  Toxin A: GMT at Day 210, 65 and older | 110.3 [72.4 to 168.1] | 151.9 [96.7 to 238.6] | 190.5 [131.4 to 276.1] | 10.4 [9.6 to 11.2]
  Toxin B: GMT at Day 0, 50 - < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  Toxin B: GMT at Day 0, 50 - < 65 | 15.4 [12.3 to 19.4] | 16.7 [13.1 to 21.3] | 19.3 [14.3 to 26.2] | 13.6 [9.3 to 19.8]
  Toxin B: GMT at Day 35, 50 - < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  Toxin B: GMT at Day 35, 50 - < 65 | 59.4 [36.6 to 96.2] | 114.2 [71.4 to 182.9] | 61.7 [37.2 to 102.4] | 14.2 [9.7 to 20.9]
  Toxin B: GMT at Day 56, 50 - < 65: number analyzed (Participants) | 67 | 68 | 70 | 22
  Toxin B: GMT at Day 56, 50 - < 65 | 56.9 [36.5 to 88.7] | 95.0 [62.5 to 144.3] | 53.9 [34.3 to 84.6] | 14.9 [10.4 to 21.4]
  Toxin B: GMT at Day 210, 50 - < 65: number analyzed (Participants) | 65 | 66 | 68 | 22
  Toxin B: GMT at Day 210, 50 - < 65 | 44.1 [29.0 to 67.0] | 69.9 [47.4 to 102.9] | 40.3 [25.6 to 63.3] | 14.1 [9.7 to 20.3]
  Toxin B: GMT at Day 0, 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  Toxin B: GMT at Day 0, 65 and older | 19.5 [14.6 to 26.0] | 15.2 [12.0 to 19.2] | 18.9 [14.1 to 25.5] | 24.1 [13.9 to 42.0]
  Toxin B: GMT at Day 35, 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  Toxin B: GMT at Day 35, 65 and older | 88.7 [52.0 to 151.4] | 86.7 [52.6 to 142.9] | 61.6 [38.9 to 97.6] | 23.8 [13.7 to 41.3]
  Toxin B: GMT at Day 56, 65 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  Toxin B: GMT at Day 56, 65 and older | 84.8 [53.5 to 134.5] | 57.9 [38.3 to 87.5] | 50.7 [32.9 to 78.2] | 23.8 [14.2 to 40.1]
  Toxin B: GMT at Day 210, 65 and older: number analyzed (Participants) | 69 | 66 | 69 | 23
  Toxin B: GMT at Day 210, 65 and older | 58.6 [38.0 to 90.3] | 53.3 [35.8 to 79.5] | 45.9 [30.2 to 69.7] | 20.9 [12.3 to 35.7]

12. Secondary Outcome: Responder Rate (RR) for Neutralizing Antibodies Against Both Toxin A and Toxin B
Description: Responder Rate (RR) (defined as percentage of subjects achieving a ≥4-fold increase in neutralizing antibody titer from Day 0) for neutralizing antibodies against both Toxin A and Toxin B on Days 35, 56, 120* and 210
  * TNA in sera from Day 120 were to be measured only if meaningful in view of the Day 56 and Day 210 results; in fact Day 120 TNA was not measured.
Time Frame: Days 35, 56, 120, 210
Population: PP210 = per protocol population defined as subjects without major protocol deviation up to Day 210
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 137 | 135 | 141 | 46
percentage of participants
  RR Day 35 | 42.3 [34.4 to 50.7] | 54.1 [45.7 to 62.3] | 40.4 [32.7 to 48.7] | 0.0 [0.0 to 7.7]
  RR Day 56 | 46.0 [37.9 to 54.3] | 51.9 [43.5 to 60.1] | 36.9 [29.4 to 45.1] | 0.0 [0.0 to 7.7]
  RR Day 210: number analyzed (Participants) | 134 | 132 | 137 | 45
  RR Day 210 | 38.1 [30.3 to 46.5] | 46.2 [37.9 to 54.7] | 27.7 [20.9 to 35.8] | 0.0 [0.0 to 7.9]

13. Secondary Outcome: Responder Rate (RR) for Toxin A Neutralizing Antibodies
Description: Responder Rate (RR) (defined as percentage of subjects achieving a ≥4-fold increase in neutralizing antibody titer from Day 0) for neutralizing antibodies against Toxin A on Days 35, 56, 120* and 210
  * TNA in sera from Day 120 were to be measured only if meaningful in view of the Day 56 and Day 210 results; in fact Day 120 TNA was not measured.
Time Frame: Days 35, 56, 120 and 210
Population: PP210 = per protocol population defined as subjects without major protocol deviation up to Day 210
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 137 | 135 | 141 | 46
percentage of participants
  RR Day 35 | 55.5 [47.1 to 63.5] | 68.1 [59.9 to 75.4] | 67.4 [59.3 to 74.6] | 0.0 [0.0 to 7.7]
  RR Day 56 | 68.6 [60.4 to 75.8] | 78.5 [70.9 to 84.6] | 76.6 [69.0 to 82.8] | 0.0 [0.0 to 7.7]
  RR Day 210: number analyzed (Participants) | 134 | 132 | 137 | 45
  RR Day 210 | 62.7 [54.3 to 70.4] | 75.0 [67.0 to 81.6] | 84.7 [77.7 to 89.8] | 0.0 [0.0 to 7.9]

14. Secondary Outcome: Responder Rate (RR) for Toxin B Neutralizing Antibodies
Description: Responder Rate (RR) (defined as percentage of subjects achieving a ≥4-fold increase in neutralizing antibody titer from Day 0) for neutralizing antibodies against Toxin B on Days 35, 56, 120* and 210
  * TNA in sera from Day 120 were to be measured only if meaningful in view of the Day 56 and Day 210 results; in fact Day 120 TNA was not measured.
Time Frame: Days 35, 56, 120 and 210
Population: PP210 = per protocol population defined as subjects without major protocol deviation up to Day 210
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 137 | 135 | 141 | 46
percentage of participants
  RR Day 35 | 48.2 [40.0 to 56.5] | 57.8 [49.3 to 65.8] | 42.6 [34.7 to 50.8] | 0.0 [0.0 to 7.7]
  RR Day 56 | 52.6 [44.2 to 60.7] | 56.3 [47.9 to 64.4] | 38.3 [30.7 to 46.5] | 0.0 [0.0 to 7.7]
  RR Day 210: number analyzed (Participants) | 134 | 132 | 137 | 45
  RR Day 210 | 39.6 [31.7 to 48.0] | 47.0 [38.7 to 55.4] | 27.7 [20.9 to 35.8] | 2.2 [0.4 to 11.6]

15. Secondary Outcome: Responder Rate (RR) for Neutralizing Antibodies Against Toxin A, Against Toxin B and Against Both Toxin A and Toxin B Stratified by Age Group
Description: Responder Rate for neutralizing antibodies against Toxin A (RR Tox A), against Toxin B (RR Tox B) and against both Toxin A and Toxin B (RR Tox A and B) on Days 35, 56, 120* and 210, stratified by age group (subjects 50 - < 65 years and 65 years and older)
  * TNA in sera from Day 120 were to be measured only if meaningful in view of the Day 56 and Day 210 results; in fact Day 120 TNA was not measured.
Time Frame: Days 35, 56, 120 and 210
Population: PP210 = per protocol population defined as subjects without major protocol deviation up to Day 210
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 137 | 135 | 141 | 46
percentage of participants
  RR Tox A and B Day 35, 50 - < 60: number analyzed (Participants) | 67 | 68 | 70 | 22
  RR Tox A and B Day 35, 50 - < 60 | 38.8 [28.0 to 50.8] | 55.9 [44.1 to 67.1] | 42.9 [31.9 to 54.5] | 0.0 [0.0 to 14.9]
  RR Tox A and B Day 56, 50 - < 60: number analyzed (Participants) | 67 | 68 | 70 | 22
  RR Tox A and B Day 56, 50 - < 60 | 49.3 [37.7 to 60.9] | 57.4 [45.5 to 68.4] | 35.7 [25.5 to 47.4] | 0.0 [0.0 to 14.9]
  RR Tox A and B Day 210, 50 - < 60: number analyzed (Participants) | 65 | 66 | 68 | 22
  RR Tox A and B Day 210, 50 - < 60 | 36.9 [26.2 to 49.1] | 50.0 [38.3 to 61.7] | 25.0 [16.2 to 36.4] | 0.0 [0.0 to 14.9]
  RR Tox A and B Day 35, 60 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  RR Tox A and B Day 35, 60 and older | 45.7 [34.6 to 57.3] | 52.2 [40.5 to 63.7] | 38.0 [27.6 to 49.7] | 0.0 [0.0 to 13.8]
  RR Tox A and B Day 56, 60 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  RR Tox A and B Day 56, 60 and older | 42.9 [31.9 to 54.5] | 46.3 [34.9 to 58.1] | 38.0 [27.6 to 49.7] | 0.0 [0.0 to 13.8]
  RR Tox A and B Day 210, 60 and older: number analyzed (Participants) | 69 | 66 | 69 | 23
  RR Tox A and B Day 210, 60 and older | 39.1 [28.5 to 50.9] | 42.4 [31.2 to 54.4] | 30.4 [20.8 to 42.1] | 0.0 [0.0 to 14.3]
  RR Tox A Day 35, 50 - < 60: number analyzed (Participants) | 67 | 68 | 70 | 22
  RR Tox A Day 35, 50 - < 60 | 53.7 [41.9 to 65.1] | 70.6 [58.9 to 80.1] | 67.1 [55.5 to 77.0] | 0.0 [0.0 to 14.9]
  RR Tox A Day 56, 50 - < 60: number analyzed (Participants) | 67 | 68 | 70 | 22
  RR Tox A Day 56, 50 - < 60 | 67.2 [55.3 to 77.2] | 77.9 [66.7 to 86.2] | 72.9 [61.5 to 81.9] | 0.0 [0.0 to 14.9]
  RR Tox A Day 210, 50 - < 60: number analyzed (Participants) | 65 | 66 | 68 | 22
  RR Tox A Day 210, 50 - < 60 | 56.9 [44.8 to 68.2] | 77.3 [65.8 to 85.7] | 83.8 [73.3 to 90.7] | 0.0 [0.0 to 14.9]
  RR Tox A Day 35, 60 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  RR Tox A Day 35, 60 and older | 57.1 [45.5 to 68.1] | 65.7 [53.7 to 75.9] | 67.6 [56.1 to 77.3] | 0.0 [0.0 to 13.8]
  RR Tox A Day 56, 60 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  RR Tox A Day 56, 60 and older | 70.0 [58.5 to 79.5] | 79.1 [67.9 to 87.1] | 80.3 [69.6 to 87.9] | 0.0 [0.0 to 13.9]
  RR Tox A Day 210, 60 and older: number analyzed (Participants) | 69 | 66 | 69 | 23
  RR Tox A Day 210, 60 and older | 68.1 [56.4 to 77.9] | 72.7 [61.0 to 82.0] | 85.5 [75.3 to 91.9] | 0.0 [0.0 to 14.3]
  RR Tox B Day 35, 50 - < 60: number analyzed (Participants) | 67 | 68 | 70 | 22
  RR Tox B Day 35, 50 - < 60 | 43.3 [32.1 to 55.2] | 61.8 [49.9 to 72.4] | 42.9 [31.9 to 54.5] | 0.0 [0.0 to 14.9]
  RR Tox B Day 56, 50 - < 60: number analyzed (Participants) | 67 | 68 | 70 | 22
  RR Tox B Day 56, 50 - < 60 | 52.2 [40.5 to 63.7] | 61.8 [49.9 to 72.4] | 37.1 [26.8 to 48.9] | 0.0 [0.0 to 14.9]
  RR Tox B Day 210, 50 - < 60: number analyzed (Participants) | 65 | 66 | 68 | 22
  RR Tox B Day 210, 50 - < 60 | 40.0 [29.0 to 52.1] | 50.0 [38.3 to 61.7] | 25.0 [16.2 to 36.4] | 4.5 [0.8 to 21.8]
  RR Tox B Day 35, 60 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  RR Tox B Day 35, 60 and older | 52.9 [41.3 to 64.1] | 53.7 [41.9 to 65.1] | 42.3 [31.5 to 53.8] | 0.0 [0.0 to 13.8]
  RR Tox B Day 56, 60 and older: number analyzed (Participants) | 70 | 67 | 71 | 24
  RR Tox B Day 56, 60 and older | 52.9 [41.3 to 64.1] | 50.7 [39.1 to 62.3] | 39.4 [28.9 to 51.1] | 0.0 [0.0 to 13.8]
  RR Tox B Day 210, 60 and older: number analyzed (Participants) | 69 | 66 | 69 | 23
  RR Tox B Day 210, 60 and older | 39.1 [28.5 to 50.9] | 43.9 [32.6 to 55.9] | 30.4 [20.8 to 42.1] | 0.0 [0.0 to 14.3]

16. Secondary Outcome: Rate of Study Participants With at Least One SAE (Serious Adverse Event)
Description: percentage of study participants with at least one SAE starting up to Day 56 and up to Day 210
Time Frame: Day 56 and Day 210
Population: Safety Population = study participants who received at least one study vaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 148 | 152 | 152 | 48
percentage of participants
  up to Day 56 | 0.7 [0.1 to 3.7] | 0.7 [0.1 to 3.6] | 0.0 [0.0 to 2.5] | 4.2 [1.2 to 14.0]
  up to Day 210 | 2.7 [1.1 to 6.7] | 3.3 [1.4 to 7.5] | 2.0 [0.7 to 5.6] | 4.2 [1.2 to 14.0]

17. Secondary Outcome: Rate of Study Participants With at Least One Related SAE
Description: percentage of study participants with at least one related SAE starting up to Day 56 and up to Day 210
Time Frame: Day 56 and Day 210
Population: Safety Population = study participants with at least one study vaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 148 | 152 | 152 | 48
percentage of participants
  up to Day 56 | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 7.4]
  up to Day 210 | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 2.5] | 0.0 [0.0 to 7.4]

18. Secondary Outcome: Rate of Study Participants With at Least One Unsolicited AEs (Adverse Event)
Description: percentage of study participants with at least one unsolicited AE starting up to Day 56 and Day 210 (incl. clinically significant laboratory parameter changes)
Time Frame: Day 56 and Day 210
Population: Safety Population = study participants with at least one study vaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 148 | 152 | 152 | 48
percentage of participants
  up to Day 56 | 33.1 [26.0 to 41.0] | 32.2 [25.3 to 40.0] | 30.9 [24.1 to 38.7] | 29.2 [18.2 to 43.2]
  up to Day 210 | 43.9 [36.2 to 52.0] | 39.5 [32.1 to 47.4] | 40.1 [32.7 to 48.1] | 37.5 [25.2 to 51.6]

19. Secondary Outcome: Rate of Study Participants With at Least One Related Unsolicited AE
Description: percentage of study participants with at least one related unsolicited AE starting up to Day 56 and Day 210 (incl. clinically significant laboratory parameter changes)
Time Frame: Day 56 and Day 210
Population: Safety Population = study participants with at least one study vaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 148 | 152 | 152 | 48
percentage of participants
  up to Day 56 | 11.5 [7.3 to 17.6] | 12.5 [8.2 to 18.7] | 7.9 [4.6 to 13.3] | 4.2 [1.2 to 14.0]
  up to Day 210 | 11.5 [7.3 to 17.6] | 13.2 [8.7 to 19.5] | 7.9 [4.6 to 13.3] | 4.2 [1.2 to 14.0]

20. Secondary Outcome: Rates of Study Participants With at Least One Solicited Local and Systemic AE
Description: percentage of study participants with solicited local and systemic AE within 7 days after each and after any vaccination, collected via a subject diary with predefined terms
Time Frame: within 7 Days after each vaccination
Population: Safety Population = study participants with at least one study vaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 148 | 152 | 152 | 48
percentage of participants
  any local solicited AE, after 1st vaccination | 17.0 [11.8 to 23.9] | 19.1 [13.6 to 26.1] | 19.7 [14.2 to 26.8] | 14.9 [7.4 to 27.7]
  any local solicited AE, after 2nd vaccination | 17.2 [12.0 to 24.2] | 29.6 [22.9 to 37.3] | 30.9 [24.1 to 38.7] | 12.8 [6.0 to 25.2]
  any local solicited AE, after 3rd vaccination | 15.3 [10.3 to 22.0] | 29.3 [22.5 to 37.1] | 25.0 [18.7 to 32.5] | 10.6 [4.6 to 22.6]
  any local solicited AE, overall | 28.6 [21.9 to 36.3] | 48.0 [40.2 to 55.9] | 46.7 [39.0 to 54.6] | 21.3 [12.0 to 34.9]
  any systemic solicited AE, after 1st vaccination | 23.1 [17.0 to 30.6] | 23.7 [17.6 to 31.0] | 21.1 [15.3 to 28.2] | 21.3 [12.0 to 34.9]
  any systemic solicited AE, after 2nd vaccination | 17.8 [12.5 to 24.8] | 27.6 [21.1 to 35.2] | 17.8 [12.5 to 24.6] | 14.9 [7.4 to 27.7]
  any systemic solicited AE, after 3rd vaccination | 13.2 [8.6 to 19.7] | 16.3 [11.2 to 23.1] | 16.9 [11.7 to 23.7] | 12.8 [6.0 to 25.2]
  any systemic solicited AE, overall | 35.4 [28.1 to 43.4] | 42.1 [34.5 to 50.1] | 37.5 [30.2 to 45.4] | 38.3 [25.8 to 52.6]

21. Secondary Outcome: Rates of Study Participants With at Least One SAE, Related SAE, Unsolicited AE and Related Unsolicited AE Stratified by Age Group
Description: percentage of study participants with at least one SAE, related SAE, unsolicited (unsol.) AE (incl. clinically significant laboratory parameter changes) and related unsolicited AE, starting up to Day 56 and Day 210, stratified by age group (subjects 50 - < 65 years and 65 years and older (65+))
Time Frame: Day 56 and Day 210
Population: Safety Population = study participants with at least one study vaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 148 | 152 | 152 | 48
percentage of participants
  SAEs up to Day 56, 50 - < 60: number analyzed (Participants) | 72 | 77 | 77 | 24
  SAEs up to Day 56, 50 - < 60 | 0.0 [0.0 to 5.1] | 1.3 [0.2 to 7.0] | 0.0 [0.0 to 4.8] | 8.3 [2.3 to 25.8]
  SAEs up to Day 210, 50 - < 60: number analyzed (Participants) | 72 | 77 | 77 | 24
  SAEs up to Day 210, 50 - < 60 | 2.8 [0.8 to 9.6] | 3.9 [1.3 to 10.8] | 0.0 [0.0 to 4.8] | 8.3 [2.3 to 25.8]
  related SAEs up to Day 56, 50 - < 60: number analyzed (Participants) | 72 | 77 | 77 | 24
  related SAEs up to Day 56, 50 - < 60 | 0.0 [0.0 to 5.1] | 0.0 [0.0 to 4.8] | 0.0 [0.0 to 4.8] | 0.0 [0.0 to 13.8]
  related SAEs up to Day 210, 50 - < 60: number analyzed (Participants) | 72 | 77 | 77 | 24
  related SAEs up to Day 210, 50 - < 60 | 0.0 [0.0 to 5.1] | 0.0 [0.0 to 4.8] | 0.0 [0.0 to 4.8] | 0.0 [0.0 to 13.8]
  any unsolicited AE up to Day 56, 50 - < 60: number analyzed (Participants) | 72 | 77 | 77 | 24
  any unsolicited AE up to Day 56, 50 - < 60 | 37.5 [27.2 to 49.0] | 33.8 [24.2 to 44.9] | 28.6 [19.7 to 39.5] | 25.0 [12.0 to 44.9]
  any unsolicited AE up to Day 210, 50 - < 60: number analyzed (Participants) | 72 | 77 | 77 | 24
  any unsolicited AE up to Day 210, 50 - < 60 | 50.0 [38.7 to 61.3] | 41.6 [31.2 to 52.7] | 39.0 [28.8 to 50.1] | 33.3 [18.0 to 53.3]
  any related unsolicited AE up to Day 56, 50 - < 60: number analyzed (Participants) | 72 | 77 | 77 | 24
  any related unsolicited AE up to Day 56, 50 - < 60 | 12.5 [6.7 to 22.1] | 11.7 [6.3 to 20.7] | 9.1 [4.5 to 17.6] | 8.3 [2.3 to 25.8]
  any related unsolicited AE up to Day 210, 50 -< 60: number analyzed (Participants) | 72 | 77 | 77 | 24
  any related unsolicited AE up to Day 210, 50 -< 60 | 12.5 [6.7 to 22.1] | 13.0 [7.2 to 22.3] | 9.1 [4.5 to 17.6] | 8.3 [2.3 to 25.8]
  SAEs up to Day 56, 65 and older: number analyzed (Participants) | 76 | 75 | 75 | 24
  SAEs up to Day 56, 65 and older | 1.3 [0.2 to 7.1] | 0.0 [0.0 to 4.9] | 0.0 [0.0 to 4.9] | 0.0 [0.0 to 13.8]
  SAEs up to Day 210, 65 and older: number analyzed (Participants) | 76 | 75 | 75 | 24
  SAEs up to Day 210, 65 and older | 2.6 [0.7 to 9.1] | 2.7 [0.7 to 9.2] | 4.0 [1.4 to 11.1] | 0.0 [0.0 to 13.8]
  related SAEs up to Day 56, 65 and older: number analyzed (Participants) | 76 | 75 | 75 | 24
  related SAEs up to Day 56, 65 and older | 0.0 [0.0 to 4.8] | 0.0 [0.0 to 4.9] | 0.0 [0.0 to 4.9] | 0.0 [0.0 to 13.8]
  related SAEs up to Day 210, 65 and older: number analyzed (Participants) | 76 | 75 | 75 | 24
  related SAEs up to Day 210, 65 and older | 0.0 [0.0 to 4.8] | 0.0 [0.0 to 4.9] | 0.0 [0.0 to 4.9] | 0.0 [0.0 to 13.8]
  any unsolicited AE up to Day 56, 60 and older: number analyzed (Participants) | 76 | 75 | 75 | 24
  any unsolicited AE up to Day 56, 60 and older | 28.9 [20.0 to 40.0] | 30.7 [21.4 to 41.8] | 33.3 [23.7 to 44.6] | 33.3 [18.0 to 53.3]
  any unsolicited AE up to Day 210, 60 and older: number analyzed (Participants) | 76 | 75 | 75 | 24
  any unsolicited AE up to Day 210, 60 and older | 38.2 [28.1 to 49.4] | 37.3 [27.3 to 48.6] | 41.3 [30.9 to 52.6] | 41.7 [24.5 to 61.2]
  any related unsol. AE up to Day 56, 60 and older: number analyzed (Participants) | 76 | 75 | 75 | 24
  any related unsol. AE up to Day 56, 60 and older | 10.5 [5.4 to 19.4] | 13.3 [7.4 to 22.8] | 6.7 [2.9 to 14.7] | 0.0 [0.0 to 13.8]
  any related unsol. AE up to Day 210, 60 and older: number analyzed (Participants) | 76 | 75 | 75 | 24
  any related unsol. AE up to Day 210, 60 and older | 10.5 [5.4 to 19.4] | 13.3 [7.4 to 22.8] | 6.7 [2.9 to 14.7] | 0.0 [0.0 to 13.8]

22. Secondary Outcome: Rates of Study Participants With at Least One Solicited Local and Systemic AE Within 7 Days After Each and Any Vaccination Stratified by Age Group
Description: percentage of participants with solicited (sol.) local and systemic AEs within 7 days after each and after any vaccination (vacc.), collected via a subject diary with predefined terms, stratified by age group (subjects 50 - < 65 years and 65 years and older)
Time Frame: within 7 Days after each vaccination
Population: Safety Population = study participants with at least one study vaccination
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Number analyzed (Participants) | 148 | 152 | 152 | 48
percentage of participants
  any local sol. AE, after 1st vacc., 50 -< 65: number analyzed (Participants) | 72 | 77 | 77 | 24
  any local sol. AE, after 1st vacc., 50 -< 65 | 18.1 [10.9 to 28.5] | 27.3 [18.6 to 38.1] | 18.2 [11.2 to 28.2] | 17.4 [7.0 to 37.1]
  any local sol. AE, after 2nd vacc., 50 -< 65: number analyzed (Participants) | 72 | 77 | 77 | 24
  any local sol. AE, after 2nd vacc., 50 -< 65 | 14.3 [7.9 to 24.3] | 31.2 [21.9 to 42.2] | 33.8 [24.2 to 44.9] | 17.4 [7.0 to 37.1]
  any local sol. AE, after 3rd vacc., 50 -< 65: number analyzed (Participants) | 72 | 77 | 77 | 24
  any local sol. AE, after 3rd vacc., 50 -< 65 | 17.4 [10.2 to 28.0] | 32.4 [22.9 to 43.7] | 23.0 [14.9 to 33.7] | 13.0 [4.5 to 32.1]
  any local sol. AE, overall, 50 -< 65: number analyzed (Participants) | 72 | 77 | 77 | 24
  any local sol. AE, overall, 50 -< 65 | 29.2 [19.9 to 40.5] | 53.2 [42.2 to 64.0] | 51.9 [41.0 to 62.7] | 21.7 [9.7 to 41.9]
  any local sol. AE, after 1st vacc., 65 and older: number analyzed (Participants) | 76 | 75 | 75 | 24
  any local sol. AE, after 1st vacc., 65 and older | 16.0 [9.4 to 25.9] | 10.7 [5.5 to 19.7] | 21.3 [13.6 to 31.9] | 12.5 [4.3 to 31.0]
  any local sol. AE, after 2nd vacc., 65 and older: number analyzed (Participants) | 76 | 75 | 75 | 24
  any local sol. AE, after 2nd vacc., 65 and older | 20.0 [12.5 to 30.4] | 28.0 [19.1 to 39.0] | 28.0 [19.1 to 39.0] | 8.3 [2.3 to 25.8]
  any local sol. AE, after 3rd vacc., 65 and older: number analyzed (Participants) | 76 | 75 | 75 | 24
  any local sol. AE, after 3rd vacc., 65 and older | 13.3 [7.4 to 22.8] | 26.0 [17.3 to 37.1] | 27.0 [18.2 to 38.1] | 8.3 [2.3 to 25.8]
  any local sol. AE, overall, 65 and older: number analyzed (Participants) | 76 | 75 | 75 | 24
  any local sol. AE, overall, 65 and older | 28.0 [19.1 to 39.0] | 42.7 [32.1 to 53.9] | 41.3 [30.9 to 52.6] | 20.8 [9.2 to 40.5]
  any systemic sol. AE, after 1st vacc., 50 - < 65: number analyzed (Participants) | 72 | 77 | 77 | 24
  any systemic sol. AE, after 1st vacc., 50 - < 65 | 29.2 [19.9 to 40.5] | 26.0 [17.5 to 36.7] | 24.7 [16.4 to 35.4] | 21.7 [9.7 to 41.9]
  any systemic sol. AE, after 2nd vacc., 50 - < 65: number analyzed (Participants) | 72 | 77 | 77 | 24
  any systemic sol. AE, after 2nd vacc., 50 - < 65 | 16.9 [9.9 to 27.3] | 28.6 [19.7 to 39.5] | 18.2 [11.2 to 28.2] | 21.7 [9.7 to 41.9]
  any systemic sol. AE, after 3rd vacc., 50 - < 65: number analyzed (Participants) | 72 | 77 | 77 | 24
  any systemic sol. AE, after 3rd vacc., 50 - < 65 | 18.8 [11.4 to 29.6] | 14.9 [8.5 to 24.7] | 21.6 [13.8 to 32.3] | 8.7 [2.4 to 26.8]
  any systemic sol. AE, overall, 50 - < 65: number analyzed (Participants) | 72 | 77 | 77 | 24
  any systemic sol. AE, overall, 50 - < 65 | 40.3 [29.7 to 51.8] | 46.8 [36.0 to 57.8] | 44.2 [33.6 to 55.3] | 39.1 [22.2 to 59.2]
  any systemic sol. AE, after 1st vacc.,65 and older: number analyzed (Participants) | 76 | 75 | 75 | 24
  any systemic sol. AE, after 1st vacc.,65 and older | 17.3 [10.4 to 27.4] | 21.3 [13.6 to 31.9] | 17.3 [10.4 to 27.4] | 20.8 [9.2 to 40.5]
  any systemic sol. AE, after 2nd vacc.,65 and older: number analyzed (Participants) | 76 | 75 | 75 | 24
  any systemic sol. AE, after 2nd vacc.,65 and older | 18.7 [11.5 to 28.9] | 26.7 [18.0 to 37.6] | 17.3 [10.4 to 27.4] | 8.3 [2.3 to 25.8]
  any systemic sol. AE, after 3rd vacc.,65 and older: number analyzed (Participants) | 76 | 75 | 75 | 24
  any systemic sol. AE, after 3rd vacc.,65 and older | 8.0 [3.7 to 16.4] | 17.8 [10.7 to 28.1] | 12.2 [6.5 to 21.5] | 16.7 [6.7 to 35.9]
  any systemic sol. AE, overall ,65 and older: number analyzed (Participants) | 76 | 75 | 75 | 24
  any systemic sol. AE, overall ,65 and older | 30.7 [21.4 to 41.8] | 37.3 [27.3 to 48.6] | 30.7 [21.4 to 41.8] | 37.5 [21.2 to 57.3]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected throughout the study, i.e., up to Day 210. Unsolicited local and systemic AEs are defined as follows: any of the solicited local or systemic AEs which has an onset date more than 6 days after vaccination OR any other symptom or untoward medical event. Additionally, subject diaries were dispensed covering the first 7 days after each vaccination (starting on the day of vaccination) to capture predefined AEs typical for vaccinations.
Description: Solicited AEs listed (predefined) in the diaries comprised injection site reactions (pain, itching, tenderness, induration (hardening), swelling, erythema (redness)) or systemic reactions (headache, muscle pain, fever (oral), flu-like symptoms, nausea, vomiting, rash, excessive fatigue). Solicited AEs are per definition regarded as related to IMP.
Arm/Group | VLA84 75 mcg (Microgram) w/o Alum | VLA84 200 mcg w/o Alum | VLA84 200 mcg With Alum | Placebo
Serious Adverse Events (participants affected / at risk) | 4/148 | 5/152 | 3/152 | 2/48
Other Adverse Events (participants affected / at risk) | 75/148 | 94/152 | 89/152 | 23/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VLA84 75 mcg (Microgram) w/o Alum (N=148) | VLA84 200 mcg w/o Alum (N=152) | VLA84 200 mcg With Alum (N=152) | Placebo (N=48)
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 1 | 0
Histoplasmosis (Infections and infestations) | 1 | 0 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Device dislocation (General disorders) | 1 | 0 | 0 | 0
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Inguinal hernia repair (Surgical and medical procedures) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VLA84 75 mcg (Microgram) w/o Alum (N=148) | VLA84 200 mcg w/o Alum (N=152) | VLA84 200 mcg With Alum (N=152) | Placebo (N=48)
Injection site pain (General disorders) | 33 | 62 | 60 | 8
Fatigue (General disorders) | 25 | 32 | 23 | 5
Influenza like illness (General disorders) | 17 | 30 | 21 | 4
Injection site erythema (General disorders) | 13 | 23 | 20 | 4
Injection site pruritus (General disorders) | 9 | 18 | 15 | 1
Injection site swelling (General disorders) | 7 | 14 | 17 | 2
Injection site induration (General disorders) | 6 | 14 | 12 | 3
Pyrexia (General disorders) | 4 | 9 | 3 | 0
Headache (Nervous system disorders) | 36 | 31 | 36 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 29 | 25 | 6
Nausea (Gastrointestinal disorders) | 16 | 12 | 14 | 6
Diarrhoea (Gastrointestinal disorders) | 9 | 8 | 5 | 2
Sinusitis (Infections and infestations) | 3 | 1 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not less than 60 days prior to the earlier of Publication or submission for Publication of any Manuscript Sponsor has to be provided with a copy of the Manuscript (unless the Manuscript is an abstract, presentation, or poster: not less than 30 days prior to the earlier of Publication or submission for Publication). Site shall delay Publication/ submission for Publication of the Manuscript, as the case may be, for an additional 120 days to allow patent applications to be filed.